CLINICAL TRIAL: NCT05697185
Title: Safety and Efficacy of Evolocumab in in Combination With Statin Therapy in Adults With Ischemic Stroke
Brief Title: Safety and Efficacy of Evolocumab in Ischemic Stroke
Acronym: SEEIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Junli Liang, Professor, Second Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-0012
Record Dates: First submitted 2023-01-15; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke | interventions — evolocumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the evolocumab plus statin therapy (Experimental): Patients with AIS are treated with atorvastatin (40mg) daily and evolocumab (420 mg) every months throughout the study period
  Interventions: Drug: Evolocumab
- the statin alone therapy (No Intervention): Patients with AIS are treated with atorvastatin (40mg) daily throughout the study period.

INTERVENTIONS:
Drug: Evolocumab — Patients were randomly assigned of the ratio of 1:1 using a computer-generated random number and divided into two treatment groups: the statin alone therapy and the evolocumab plus statin therapy.
  Arms: the evolocumab plus statin therapy

SUMMARY:
The goal of this clinical trial is to evaluate the effect of evolocumab in combination with statin therapy (atorvastatin) in acute ischemic stroke (AIS).

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18-80 years
2. Time of onset: within 1 week
3. NIHSS score ≤12
4. Acute ischemic stroke confirmed by head CT or MRI
5. Premorbid mRS ≤1
6. Signed informed consent

Exclusion Criteria:

1. Intracranial hemorrhage found by head CT
2. Severe hepatic or renal dysfunction
3. Pregnant females
4. Abnormal elevation of creatine phosphokinase
5. Blood sugar is out of control
6. Receiving statins within 1 month before onset
7. Not willing and able to comply with scheduled visits, lifestyle guidelines, treatment plan, laboratory tests, and other study procedures
8. Unsuitable for this clinical studies assessed by researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in LDL-C | baseline, 4 weeks, 8 weeks, 12 weeks after treatment

SECONDARY OUTCOMES:
Vascular events | 3 months, 6months
  incidence of Transient ischemic attack, stroke or other vascular events
mRS (0-2) | 3 months, 6months
  proportion of mRS (0-2)
death of any causes | 12 months
  proportion of death

CONTACTS AND LOCATIONS:
Overall Officials: Junli Liang, PhD, Study Director — The Second Affiliated Hospital of Guangxi Medical University, Nanning, China

REFERENCES:
- [Derived] Qiu X, Liang Y, Wei Y, Lu M, Mei Y, Tang S, Tang J, Liang J, Liang J. Evolocumab for early reduction of LDL-C levels in patients with acute ischemic stroke: a randomized controlled trial. Front Neurol. 2024 Dec 23;15:1454608. doi: 10.3389/fneur.2024.1454608. eCollection 2024. PMID 39764289